CLINICAL TRIAL: NCT01511900
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of CAT-1004 in Patients With Type 2 Diabetes
Brief Title: A Multiple Ascending Dose Study of CAT-1004 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Catabasis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: CAT 1004 102
Record Dates: First submitted 2012-01-08; First posted 2012-01-19 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1: Dose level 1 (Experimental): Multiple dose orally: CAT-1004 Dose level 1 or placebo
  Interventions: Drug: CAT 1004; Drug: Placebo
- Cohort 2: Dose level 2 (Experimental): Multiple dose orally: CAT-1004 Dose level 2 or placebo
  Interventions: Drug: Placebo; Drug: CAT 1004
- Cohort 3: Dose level 3 (Experimental): Multiple dose orally: CAT-1004 Dose level 3 or placebo
  Interventions: Drug: Placebo; Drug: CAT 1004
- Cohort 4: Dose level 4 (Experimental): Multiple dose orally: CAT-1004 Dose level 4 or placebo
  Interventions: Drug: Placebo; Drug: CAT 1004
- Cohort 5: Dose level TBD (Experimental): Multiple dose orally: CAT-1004 Dose level TBD or placebo
  Interventions: Drug: Placebo; Drug: CAT 1004

INTERVENTIONS:
Drug: CAT 1004 — Multiple dose oral administration once daily for 14 days of CAT 1004 at dose level 1-9 subjects will be treated with CAT-1004
  Arms: Cohort 1: Dose level 1
Drug: Placebo — Multiple dose oral administration of placebo daily for 14 days-3 subjects will be treated with placebo per cohort
Drug: CAT 1004 — Multiple dose oral administration once daily for 14 days of CAT 1004 at dose level 2 -9 subjects will be treated with CAT-1004
  Arms: Cohort 2: Dose level 2
Drug: CAT 1004 — Multiple dose oral administration BID for 14 days of CAT 1004 at dose level 3-9 subjects will be treated with CAT-1004
  Arms: Cohort 3: Dose level 3
Drug: CAT 1004 — Multiple dose oral administration BID for 14 days of CAT 1004 at dose level 4-9 subjects will be treated with CAT-1004
  Arms: Cohort 4: Dose level 4
Drug: CAT 1004 — Multiple dose oral administration daily for 14 days of CAT 1004 at dose level TBD-9 subjects will be treated with CAT-1004
  Arms: Cohort 5: Dose level TBD

SUMMARY:
The primary objective of the study is to evaluate the safety of escalating multiple doses over 2 weeks of CAT 1004 compared to placebo in patients with Type 2 diabetes (T2D).

Secondary objectives include evaluation of the pharmacokinetics (PK) and pharmacodynamics of escalating multiple doses of CAT-1004 in patients with T2D.

ELIGIBILITY:
Inclusion Criteria:

A patient must meet all of the following criteria to be in the study:

* Age between 18 to 65 years inclusive at Screening.
* Diagnosis of T2D:
* For Part I:

  * Treated with any diet and exercise, with or without metformin (stable for ≥ 2 months).
  * HbA1c ≥ 7.0% and ≤ 10.0% if on diet and exercise alone, or ≥6.5 % and ≤ 9.0% if on metformin.
* For Part II:

  • Stable on metformin for ≥ 2 months with HbA1c ≥ 7.0% and ≤ 10.0%.
* Satisfies one of the following:

  * Females not of childbearing potential: non-pregnant and non-lactating; surgically sterile or postmenopausal for 2 years or at least 1 year with a follicle stimulating hormone assessment (FSH) greater than or equal to 40 IU/L; OR
  * Males: surgically sterile, abstinent, or patient or partner is utilizing an acceptable contraceptive method during and 3 months after the last study dose.
* On a stable diet with body mass index (BMI): 25 to 40 kg/m2 inclusive at Screening with weight stable (± 4 kg) for > 6 weeks prior to Screening.

Exclusion Criteria:

A patient will not be eligible if any of the following criteria apply:

* Use of prescription medications other than allowed medications within 30 days of planned admission to the clinic. Allowed medications include metformin, anti-hypertensives, lipid-lowering medications, thyroid replacement therapy, low-dose aspirin (81 mg/day), proton pump inhibitors and anti-depressants. Prescribed doses of these medications must have been stable for 2 months at the time of first dose.
* Clinically significant abnormalities in physical examination or vital signs at screening
* Clinically significant electrocardiogram (ECG) abnormalities as assessed by the investigator.
* Clinically significant laboratory result as assessed by the Investigator.
* The patient has a history of clinically significant medical disease including significant allergies (except for untreated, asymptomatic seasonal allergies at the time of dosing), or hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease, other than T2D, hypertension, dyslipidemia, hypothyroidism or depression.
* History or presence of malignancy within the past 5 years.
* History of Type 1 diabetes or clinically significant cardiovascular disease (including a history of unstable angina, acute myocardial infarction, coronary artery bypass graft, percutaneous coronary intervention, or New York Heart Association Class III or IV congestive heart failure within 6 months prior to screening) or clinically significant renal disease.
* History of alcohol or substance abuse or eating disorder within 2 years, OR regular use of alcohol within 6 months (>14 units of alcohol per week; 1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol).
* Use of any investigational drug or participation in any investigational study within 30 days prior to screening or 5 half-lives of the study agent, whichever is longer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of adverse events | Screening to Follow-up (Day 25)

SECONDARY OUTCOMES:
AUCinf of CAT-1004 | Days 1, 7 and 14
Glucose area under the curve for 0-24 hrs/24 and 0-4 hrs/4 | Day -2 through f/u (Day 25)
Cmax of CAT-1004 | Days 1, 7 and 14
Changes from baseline for hematology, chemistry, coagulation and urinalysis | Baseline through End of study (Day 25)
Changes from baseline for Physical exams | Baseline through end of study (Day 25)
Changes from baseline for ECGs | Baseline through end of study (Day 25)
Changes from baseline in vital signs | Baseline through end of study (Day 25)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Donovan, M.D., PhD, Study Director — Catabasis
Locations (1):
- Chula Vista, California, United States